CLINICAL TRIAL: NCT06604962
Title: Intramuscular Electrical Stimulation Using Inverse Electrodes Placement on Electromyographic Activity and Pressure Pain Threshold in the Upper Trapezius With Trigger Points - A Randomized Controlled Trial
Brief Title: Intramuscular Electrical Stimulation on Upper Trapezius With Trigger Points
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulf Medical University (Other)
Collaborators: Universidade do Sul de Santa Catarina (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-COHS-FAC-28-OCT-2023
Record Dates: First submitted 2024-09-14; First posted 2024-09-20 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Myofacial Pain Syndrome
Keywords: Myofascial trigger points; Electrical stimulation; Pressure pain threshold; Electromyography; Intramuscular stimulation; Intramuscular electrical stimulation
MeSH Terms: conditions — Facial Neuralgia

STUDY DESIGN:
Intervention Model Description: This is an experimental study to study the effects of intramuscular electrical stimulation using different electrode placements over sham comparator group
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Each random number concealed within the small opaque envelope, later all numbers concealed within the large opaque envelope. An independent researcher who was not part of the study generated 36 random (computer generated) numbers, and an office clerk was involved in the allotment of the specified interventions. The intervention provider, outcome assessors and statistician are blinded to interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I: IMES using IEP (Experimental): Participants in this group has allocated to the Intramuscular electrical stimulation using inverse electrode placement
  Interventions: Procedure: IMES using IEP
- Group II: IMES using CEP (Active Comparator): Participants in this group has allocated to the Intramuscular electrical stimulation using conventional electrode placement
  Interventions: Procedure: IMES using CEP
- Group III: Sham-IMES (Sham Comparator): Participants in this group has allocated to the Sham Intramuscular electrical stimulation
  Interventions: Other: Sham-IMES

INTERVENTIONS:
Procedure: IMES using IEP — First group (n=12) received IMES using inverse electrode placement. The needle electrode inserted into the paraspinal region was connected to the active or cathode pole of the electrical stimulator. The reference or anode pole of the electrical stimulator was connected to the electrode that was inserted into the MTrP area of the UT muscle. The muscle was stimulated for 10 min with a tolerable intensity in a single session to induce muscle relaxation
  Arms: Group I: IMES using IEP
Procedure: IMES using CEP — Second group (n=12) underwent IMES with conventional electrode placement. In this group, the cathode pole of the stimulator was connected to the needle inserted into the UT muscle, and the anode pole was connected to the needles of the paraspinal region of the cervical spine. Needle electrodes were connected using alligator clip connectors. The muscle was stimulated for 10 min with a tolerable intensity in a single session to induce muscle relaxation.
  Arms: Group II: IMES using CEP
Other: Sham-IMES — Third group (n=12) received sham-IMES. Similar to the experimental intervention groups, the cathode pole of the stimulator was connected to the needle inserted into the UT muscle, and the anode pole was connected to the needles of the paraspinal region of the cervical spine. However, the delivered IMES was very minimal intensity
  Arms: Group III: Sham-IMES

SUMMARY:
The prevalence of myofascial pain ranges from 30 to 93% and can result in sensorimotor and autonomic deficits. In routine neuromuscular electrical stimulation, conventional electrode placement (CEP) and inverse electrode placement (IEP) are used to deliver electrical stimulation for pain modulation. However, Whether pain modulation can be achieved better from the intramuscular electrical stimulation (IMES) using the inverse electrode placement (IEP) or the conventional electrode placement (CEP) is still an open issue. Thus, current study's aim to compare the effects of IMES using IEP and CEP, and sham-IMES on pressure pain threshold (PPT), EMG activity, upper trapezius (UT) muscle length and pain severity in the UT muscle with myofascial trigger points (MTrPs) among young adults.

DETAILED DESCRIPTION:
Myofascial trigger points (MTrPs) are defined as discrete areas of tenderness in taut bands of skeletal muscles that are painful. The upper trapezius (UT) muscle has been found to be often affected by MTrPs, which can result in altered sensory-motor function.

MTrPs may be related to pressure pain sensitivity and alterations in the upper trapezius muscle activity. A reduction in PPTs and increased electromyographic (EMG) activity of the UT muscle with MTrPs can be respectively interpreted as increased pain receptors sensitization and motor endplate activity.

In routine clinical practice, exercises, TrP injections, medications, and alternative therapies such as acupuncture dry needling (DN) are used to treat MTrPs. In recent years, some studies have reported that intramuscularly delivered electrical stimulation is a potential resource for the management of myofascial pain syndrome (MPS). Evidence from the literature suggests that IMES is effective in conditions such as adhesive capsulitis, MPS, and other non-traumatic musculoskeletal disorders.

In routine neuromuscular electrical stimulation, conventional electrode placement (CEP) is used, in which an active cathode pole is placed in the peripheral target tissue and a reference anode is placed over the spinal level for peripheral pain modulation. Inverse electrode placement (IEP) is a alternate electrode placement method in which a cathode pole is placed over the spinal level and an anode pole over the distal parts of the limbs. IEP model experiments on MPS and non-traumatic shoulder pain disorders achieved significant clinical outcomes for shoulder pain and associated functional disabilities.

Although IMES is effective in reducing the pain threshold and changing EMG activity, the difference between the effects of IMES based on IEP and CEP on PPT and EMG activity (%MVIC) remains unknown. In line with previous study findings, this study hypothesized that IMES using IEP would achieve significant changes in the PPT, EMG activity, muscle length, and pain severity of the UT muscle with TrPs compared with IMES using CEP and Sham-IMES

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of myofascial trigger points in the upper trapezius (UT) muscle.
* Pressure pain threshold range between 0.5 to 1.5 kg/cm2

Exclusion Criteria:

* Shoulder conditions such as adhesive capsulitis, impingement syndrome, etc.
* Individuals with cervical radiculopathy,
* Nutritional deficiencies,
* Metabolic disorders such as obesity, diabetes mellitus,
* Participation in strength training,
* Cardiac pacemakers,
* History of migraine, epilepsy, electrophobia, needle phobia, skin diseases.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-10-28 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-04-25 (Actual)

PRIMARY OUTCOMES:
Pressure pain threshold (PPT) | Day one before the treatment, day one post treatment and day three follow-up
  Pressure algometry, a device that applies an increasing force over a limited constant surface, allows the quantification of the minimum pressure, which induces pain or discomfort, indicated as the PPT. PPT in the UT muscle area was assessed using a pressure algometer (JTECH Medical Commander Echo-Algometer with Console, Serial No-0d219167) by an experienced physiotherapist blinded to the intervention groups
Upper trapezius' Surface Electromyographic activity | Day one before the treatment, day one post treatment and day three follow-up
  The surface Electromyography (EMG) recording during the experimental condition and Maximum Voluntary Isometric Contraction (MVIC) of the UT muscle was performed using a BTS FREEEMG 1000 system (BTS Bioengineering, Milan, Italy) in three sessions: day one before and after treatment and day three follow-up. EMG data collected during the MVIC of the right-side UT muscle was used as a reference value to normalize the EMG activity of the experimental condition.

SECONDARY OUTCOMES:
Pain severity | Day one before the treatment, day one post treatment and day three follow-up
  The severity of Upper Trapezius muscle pain was assessed using a visual analog scale (VAS: 0-10 cm, where 0 indicates no pain and 10 indicates severe pain), which has high intra- and inter-rater reliability to measure pain severity.
Upper trapezius' muscle length | Day one before the treatment, day one post treatment and day three follow-up
  The upper trapezius length test was used to assess the UT muscle length. This involves gently lifting the patient's head off the table, flexing the neck slightly to take the upper trapezius to a lengthened position, and assessing the range of motion and any restrictions or discomfort experienced by the patient during this maneuver. This test is a valid assessment tool for identifying restrictions or tightness in the upper trapezius muscle. The reliability coefficients for muscle length were generally higher for the healthy group compared to the neck pain group, with ICC values ranging from 0.19 to 0.93 for the neck pain group and 0.40 to 0.93 for the healthy group

CONTACTS AND LOCATIONS:
Overall Officials: Ramprasad Muthukrishnan, PhD, Study Chair — Gulf Medical University
Locations (1):
- Gulf Medical University, Ajman, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shanmugam S. Inverse Electrode Placement May Help to Improve Electrotherapeutic Effects in the Field of Chronic Pain Management. Korean J Pain. 2016 Jul;29(3):202-4. doi: 10.3344/kjp.2016.29.3.202. Epub 2016 Jul 1. No abstract available. PMID 27413488
- [Background] Shanmugam S, Mathias L, Thakur A, Kumar D. Effects of Intramuscular Electrical Stimulation Using Inversely Placed Electrodes on Myofascial Pain Syndrome in the Shoulder: A Case Series. Korean J Pain. 2016 Apr;29(2):136-40. doi: 10.3344/kjp.2016.29.2.136. Epub 2016 Apr 1. PMID 27103970
- [Background] Shanmugam S, Mathias L, Manickaraj N, Kumar KUD, Kandakurti PK, Dorairaj SK, Muthukrishnan R. Intramuscular Electrical Stimulation Combined with Therapeutic Exercises in Patients with Shoulder Adhesive Capsulitis: A Randomised Controlled Trial. Int J Surg Protoc. 2021 May 18;25(1):71-83. doi: 10.29337/ijsp.25. PMID 34056148